CLINICAL TRIAL: NCT01018758
Title: Phase II Study With Palonosetron Alone in Preventing Chemotherapy-induced Nausea and Vomiting in Untreated Patients With Aggressive Non Hodgkin's Lymphomas Who Underwent Moderately Emetogenic Chemotherapy
Brief Title: Study With Palonosetron Alone in Preventing Chemotherapy-induced Nausea and Vomiting in Untreated Patients With Aggressive Non Hodgkin's Lymphomas Who Underwent Moderately Emetogenic Chemotherapy
Acronym: NHLPal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Studio Linfomi (Other)
Responsible Party: Nicola Di Renzo, Gruppo Italiano Studio Linfomi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NHLPal
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting; Non Hodgkin's Lymphoma
Keywords: Non-Hodgkin's lymphoma; Quality of life; Chemotherapy toxicity; aggressive Non Hodgkin's Lymphomas treated with moderately emetogenic chemotherapy
MeSH Terms: conditions — Vomiting; Lymphoma, Non-Hodgkin | interventions — Palonosetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- palonosetron (Experimental)
  Interventions: Drug: Palonosetron

INTERVENTIONS:
Drug: Palonosetron — Palonosetron will be given as an intravenous bolus at the dose of 250 micrograms over 30 seconds beginning 30 minutes before chemotherapy.

SUMMARY:
This is an open-label, multicenter phase II study in patients with aggressive Non Hodgkin Lymphoma scheduled to receive moderately emetogenic polychemotherapy (according to modified Hesketh classification for antiemetic therapy).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, >18 years of age;
* Histologically or cytologically confirmed aggressive NHL (any stage in accordance with the REAL Classification);
* Patients candidates to a initial chemotherapy treatment;
* ECOG performance status of 0-1;
* Scheduled to receive a single intravenous dose of at least one of the moderately emetogenic agents (according to the modified Hesketh classification) on Day 1;
* Written informed consent;
* Female of childbearing potential must be using reliable contraceptive measures;
* Acceptable hepatic and renal functions;
* Willing and able to complete the patient diary.

Exclusion Criteria:

* Highly emetogenic chemotherapy (containing cisplatin, mechlorethamine, streptozotocin, cyclophosphamide >1500 mg/sqm; carmustine; dacarbazine; hexamethylmelamine; procarbazine), or single-agent chemotherapy with drugs having low/minimal emetogenic potential according to the Hesketh classification);
* Diagnosis of Hodgkin's Disease or Leukemia;
* Candidates to High-Dose Chemotherapy or Bone Marrow/Peripheral Blood Stem Cells Transplantation;
* Chemotherapy schedules considering the administration of emetogenic drugs in more than two consecutive days;
* Have received any investigational drugs within 30 days before study entry;
* Have received any drug with potential anti-emetic efficacy (with the exception of specific corticosteroids foreseen in the chemotherapy combination) within 24 hours of treatment initiation);
* Prior treatment with Palonosetron;
* Have a seizure disorder requiring anticonvulsant medication unless clinically stable and free of seizure activity;
* Experienced or ongoing vomiting or nausea from any organic etiology, in the screening phase;
* Clinical evidence of current or impending bowel obstruction, peritonitis, infection, uremia, severe mucositis;
* Clinically relevant electrolyte abnormalities;
* Have a known hypersensitivity to 5HT3 receptor antagonists;
* Radiotherapy within 30 days before chemotherapy administration, or scheduled to receive radiotherapy within two weeks after chemotherapy;
* Female patients who are pregnant or breast feeding;
* Inability to understand or cooperate with the study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2006-07; Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
overall rate of patients achieving a complete response (defined as no emetic episode and no use of rescue medication) | 0-120 hours

SECONDARY OUTCOMES:
rate of Complete Response | within the first 24 h after chemotherapy and 24-120 h
number of emetic episodes | within the first 24 h after chemotherapy and 24-120 h
presence of nausea graded according to Likert scale | within the first 24 h after chemotherapy and 24-120 h
time to treatment failure (first emetic episode or first need of rescue medication, whichever occurs first) | within the first 24 h after chemotherapy and 24-120 h
patient global satisfaction with antiemetic therapy, as measured by a visual analog scale (VAS) | within the first 24 h after chemotherapy and 24-120 h
toxic effects of Palonosetron | within the first 24 h after chemotherapy and 24-120 h

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Di Renzo, MD, Principal Investigator — Gruppo Italiano Studio Linfomi
Locations (1):
- Gruppo Italiano Studio Linfomi, Modena, Italy